CLINICAL TRIAL: NCT02661464
Title: A Multi-country, Prospective, Clinical Safety Study of Subjects Exposed to the Candidate Ebola Vaccines Ad26.ZEBOV and/or MVA-BN-Filo
Brief Title: Long-term Safety Follow-up of Participants Exposed to the Candidate Ebola Vaccines Ad26.ZEBOV and/or MVA-BN-Filo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the pandemic with only one participant in follow up, as the impact on the safety was determined to be negligible, the study was terminated early.
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR108112; 2015-004139-11 (EudraCT Number); VAC52150EBL4001 (Other: Janssen Vaccines & Prevention B.V.); NCT02967003 (obsolete NCT alias)
Record Dates: First submitted 2016-01-08; First posted 2016-01-22 (Estimated); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Healthy; Ebola viruses; Ebola virus disease (EVD); Filoviruses; Safety; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN Filo); Hemorrhagic fever
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exposed to Ad26.ZEBOV and/or MVA-BN Filo (Experimental): Safety Data will be collected from participants who received Ad26.ZEBOV and/or MVA-BN-Filo in Phase 1, 2 or 3 clinical studies in 6-month intervals up to 60 months after prime vaccination, including the duration in the participant's original study (Cohort 1). Female participants who became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV will be followed to the end of their pregnancy for pregnancy outcomes (Cohort 2). After the end of pregnancy, female participants will continue to be followed in Cohort 1. Safety Data for live born children to female participants will be followed up to 60 months after birth (Cohort 3).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo

INTERVENTIONS:
Biological: Ad26.ZEBOV — No vaccine will be administered in the current study. Safety data will be collected from participants who were previously exposed to Ad26.ZEBOV vaccine in Phase 1, 2, or 3 clinical studies up to 60 months and also safety data will be collected from live born children to female participants up to 60 months after birth.
Biological: MVA-BN-Filo — No vaccine will be administered in the current study. Safety data will be collected from participants who were previously exposed to MVA-BN-Filo vaccine in Phase 1, 2, or 3 clinical studies up to 60 months and also safety data will be collected from live born children to female participants up to 60 months after birth.

SUMMARY:
The purpose of the study is to assess the long-term safety profile of Ad26.ZEBOV and MVA-BN-Filo in participants previously exposed to these vaccines in Phase 1, 2, or 3 clinical studies.

DETAILED DESCRIPTION:
This is a multi-country, prospective, long-term clinical safety study for collection of serious adverse events and pregnancy outcomes following administration of Ad26.ZEBOV and/or MVA-BN-Filo vaccines among participants who were enrolled in Phase 1, 2 or 3 clinical studies. The safety data will be collected in 3 cohorts; Cohort 1- adult and pediatric participants that received Ad26.ZEBOV and/or MVA-BN-Filo in Phase 1, 2 or 3 clinical studies (adults, adolescents and children), Cohort 2- Female participants who became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV will be followed to the end of their pregnancy for pregnancy outcomes (Cohort 2). After the end of pregnancy, female participants will continue to be followed in Cohort 1. Cohort 3 - children born to female participants exposed to Ad26.ZEBOV and/or MVA-BN-Filo who became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV. Safety data will be collected on all consenting participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who participated in a Phase 1, 2 or 3 clinical study with Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV) and/or Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN-Filo) and has been exposed to Ad26.ZEBOV and/or MVA-BN-Filo (Cohort 1)
* Female who participated in a Phase 1, 2 or 3 clinical study with Ad26.ZEBOV and/or MVA-BN-Filo and became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV (Cohort 2)
* Child born to female participants exposed to Ad26.ZEBOV and/or MVA-BN-Filo in a Phase 1, 2, or 3 clinical study who became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV (Cohort 3)
* Must sign an informed consent form for the current study (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study (or let their child participate); Assent is also required of children capable of understanding the nature of the study (typically 7 years of age and older)

Exclusion Criteria:

* No exclusions beyond those that are not meeting the inclusion criteria

Ages: 0 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (16):
- Rockville, Maryland, United States
- Burkina Faso (2):
  - BoboDioulasso
  - Ouagadougou
- France (7):
  - Créteil
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Etienne
  - Strasbourg
  - Tours
- Nairobi, Kenya
- Mwanza, Tanzania
- Uganda (2):
  - Entebbe
  - Kampala
- United Kingdom (2):
  - London
  - Oxford

REFERENCES:
- [Derived] Puri A, Pollard AJ, Schmidt-Mutter C, Laine F, PrayGod G, Kibuuka H, Barry H, Nicolas JF, Lelievre JD, Sirima SB, Kamala B, Manno D, Watson-Jones D, Gaddah A, Keshinro B, Luhn K, Robinson C, Douoguih M; EBL4001 Study Group. Long-Term Clinical Safety of the Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: A Prospective, Multi-Country, Observational Study. Vaccines (Basel). 2024 Feb 17;12(2):210. doi: 10.3390/vaccines12020210. PMID 38400193

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As none of the participants met Cohort 2 eligibility criteria pre-specified in the protocol, therefore no participants were enrolled in Cohort 2. So the results were only presented for Cohorts 1 and 3.
Groups:
- Cohort 1: Ad26.ZEBOV + MVA-BN-Filo: Male or female participants who received adenovirus serotype 26 encoding the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) vaccine and/or Modified Vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo) in a Phase 1, 2 or 3 (NCT02313077, NCT02325050, NCT02376426, NCT02376400, NCT02416453, NCT02564523, NCT02543567, NCT02543268) clinical study of Ad26.ZEBOV and/or MVA-BN-Filo were enrolled in this study. Participants did not receive any vaccination in the current study. Participants were followed up for safety up to 60 months after Day 1 of vaccination (including participant's original study duration).
- Cohort 1: Placebo: Male or female participants who received placebo matching to Ad26.ZEBOV and/or MVA-BN-Filo in a Phase 1, 2 or 3 (NCT02313077, NCT02325050, NCT02376426, NCT02376400, NCT02416453, NCT02564523, NCT02543567, NCT02543268) clinical study of Ad26.ZEBOV and/or MVA-BN-Filo were enrolled in this study. Participants did not receive any vaccination in the current study. Participants were followed up for safety up to 60 months after Day 1 of vaccination (including participant's original study duration).
- Cohort 3: Ad26.ZEBOV + MVA-BN-Filo: Children born to female participants who received Ad26.ZEBOV and/or MVA-BN-Filo in a Phase 1, 2, or 3 (NCT02313077, NCT02325050, NCT02376426, NCT02376400, NCT02416453, NCT02564523, NCT02543567, NCT02543268) clinical study of Ad26.ZEBOV and/or MVA-BN-Filo and became pregnant with estimated conception within 28 days after vaccination with MVA-BN-Filo or within 3 months after vaccination with Ad26.ZEBOV in a Phase 1, 2, or 3 clinical study were enrolled in this study. Participants did not receive any vaccination in the current study. Participants were followed up for safety up to 60 months after birth.
- Cohort 3: Placebo: Children born to female participants who received placebo matching to Ad26.ZEBOV and/or MVA-BN-Filo in a Phase 1, 2, or 3 (NCT02313077, NCT02325050, NCT02376426, NCT02376400, NCT02416453, NCT02564523, NCT02543567, NCT02543268) clinical study of Ad26.ZEBOV and/or MVA-BN-Filo and became pregnant with estimated conception within 28 days after vaccination with placebo matching to MVA-BN-Filo or within 3 months after vaccination with placebo matching to Ad26.ZEBOV in a Phase 1, 2, or 3 clinical study were enrolled in this study. Participants did not receive any vaccination in the current study. Participants were followed up for safety up to 60 months after birth.
Period: Overall Study
Arm/Group | Cohort 1: Ad26.ZEBOV + MVA-BN-Filo | Cohort 1: Placebo | Cohort 3: Ad26.ZEBOV + MVA-BN-Filo | Cohort 3: Placebo
Started | 617 | 57 | 2 | 1
Full Analysis Set | 614 | 53 | 2 | 1
Completed | 295 | 0 | 1 | 0
Not Completed | 322 | 57 | 1 | 1
Not completed — Lost to Follow-up | 28 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Participants terminated prematurely | 288 | 52 | 1 | 1
Not completed — Participants who had no post-baseline visits. | 3 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were enrolled in this study and had at least one post-baseline visit, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ad26.ZEBOV + MVA-BN-Filo | Cohort 1: Placebo | Cohort 3: Ad26.ZEBOV + MVA-BN-Filo | Cohort 3: Placebo | Total
Number analyzed (Participants) | 614 | 53 | 2 | 1 | 670
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (13) | 37 (13.44) | 1.2 (0.41) | 1.3 (NA) — There was only 1 participant in the arm, hence the standard deviation could not be calculated. | 35.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 24 | 1 | 0 | 279
  Male | 360 | 29 | 1 | 1 | 391
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 4 | 0 | 0 | 39
  Not Hispanic or Latino | 569 | 46 | 2 | 1 | 618
  Unknown or Not Reported | 10 | 3 | 0 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 8 | 3 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 249 | 20 | 2 | 1 | 272
  White | 345 | 28 | 0 | 0 | 373
  More than one race | 8 | 1 | 0 | 0 | 9
  Unknown or Not Reported | 4 | 0 | 0 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  BURKINA FASO | 68 | 11 | 0 | 0 | 79
  FRANCE | 139 | 18 | 0 | 0 | 157
  KENYA | 56 | 0 | 0 | 0 | 56
  TANZANIA, UNITED REPUBLIC OF | 16 | 0 | 0 | 0 | 16
  UGANDA | 25 | 0 | 2 | 1 | 28
  UNITED KINGDOM | 170 | 10 | 0 | 0 | 180
  UNITED STATES OF AMERICA | 140 | 14 | 0 | 0 | 154

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 3: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 60 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV + MVA-BN-Filo | Cohort 1: Placebo | Cohort 3: Ad26.ZEBOV + MVA-BN-Filo | Cohort 3: Placebo
Number analyzed (Participants) | 614 | 53 | 2 | 1
Participants | 49 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Cohorts 1 and 3: Up to 60 months
Description: FAS included all participants who were enrolled in this study and had at least one post-baseline visit, regardless of the occurrence of protocol deviations. As per planned analysis of this study, the objective of this study was to collect only serious adverse events (SAEs) and other adverse events (Non-serious AEs) were not collected and analyzed in this study, hence only SAEs have been reported and presented in this study.
Arm/Group | Cohort 1: Ad26.ZEBOV + MVA-BN-Filo | Cohort 1: Placebo | Cohort 3: Ad26.ZEBOV + MVA-BN-Filo | Cohort 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/614 | 0/53 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 49/614 | 1/53 | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.ZEBOV + MVA-BN-Filo (N=614) | Cohort 1: Placebo (N=53) | Cohort 3: Ad26.ZEBOV + MVA-BN-Filo (N=2) | Cohort 3: Placebo (N=1)
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Medical Device Discomfort (General disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Food Allergy (Immune system disorders) | 1 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 3 | 0 | 2 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Typhoid Fever (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid Artery Dissection (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral Venous Thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Meningism (Nervous system disorders) | 1 | 0 | 0 | 0
Miller Fisher Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Small Fibre Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Caesarean Section (Surgical and medical procedures) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
As none of the participants met Cohort 2 eligibility criteria pre-specified in the protocol, therefore no participants were enrolled in Cohort 2. So the results were only presented for Cohorts 1 and 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02661464/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02661464/SAP_001.pdf